CLINICAL TRIAL: NCT00695175
Title: Profile of Hypertensive Patients Seen in Private Cardiology Consultation
Brief Title: National Survey on Hypertension in Cardiologic Private Practice
Acronym: Prophyl C
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Alain Castaigne, Medical Director, AstraZeneca Pharmaceuticals
Other Study IDs: NIS-CFR-DUM-2007/6
Record Dates: First submitted 2008-06-09; First posted 2008-06-11 (Estimated); Last update posted 2009-08-06 (Estimated); Status verified 2009-08

CONDITIONS: Hypertension
Keywords: Hypertension; Private cardiology consultation; Patients with hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
To evaluate (with sufficient accuracy) the profile(demographic and clinical characteristics, health care management) of hypertensive patients seen in private cardiology consultation by holding account of type of exercise of the cardiologist (private exclusive or mixed hospital and private).

ELIGIBILITY:
Inclusion Criteria:

* male or female > or = 18 years old
* Known hypertension
* agree to take part in this study

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: First three consecutive patients with hypertension seen by Cardiologists
Sampling Method: Probability Sample
Enrollment: 1800 (Actual)
Dates: Start 2008-02; Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Demographic, clinical and health care characteristics | Once

CONTACTS AND LOCATIONS:
Overall Officials: Alain Castaigne, Medical Director, Study Director — AstraZeneca
Locations (408):
- France (408):
  - Research Site, Abbeville
  - Research Site, Aire-sur-l'Adour
  - Research Site, Aix-en-Provence
  - Research Site, Aix-les-Bains
  - Research Site, Ajaccio
  - Research Site, Albert
  - Research Site, Albi
  - Research Site, Alençon
  - Research Site, Alès
  - Research Site, Ambérieu-en-Bugey
  - Research Site, Amboise
  - Research Site, Amiens
  - Research Site, Andrézieux-Bouthéon
  - Research Site, Angers
  - Research Site, Angoulême
  - Research Site, Annecy
  - Research Site, Annemasse
  - Research Site, Antibes
  - Research Site, Antony
  - Research Site, Apt
  - Research Site, Arès
  - Research Site, Argenteuil
  - Research Site, Arles
  - Research Site, Armentières
  - Research Site, Arras
  - Research Site, Asnières-sur-Seine
  - Research Site, Aubagne
  - Research Site, Aubenas
  - Research Site, Auchel
  - Research Site, Audincourt
  - Research Site, Aulnay-sous-Bois
  - Research Site, Aurillac
  - Research Site, Avignon
  - Research Site, Bagneux
  - Research Site, Bagnères-de-Bigorre
  - Research Site, Bailleul
  - Research Site, Balma
  - Research Site, Bastia
  - Research Site, Baume-les-Dames
  - Research Site, Bayeux
  - Research Site, Bayonne
  - Research Site, Beauchamp
  - Research Site, Beaumont
  - Research Site, Beaumont-de-Lomagne
  - Research Site, Beausoleil
  - Research Site, Beauvais
  - Research Site, Belfort
  - Research Site, Bellegarde-sur-Valserine
  - Research Site, Belley
  - Research Site, Bergerac
  - Research Site, Besançon
  - Research Site, Betton
  - Research Site, Bègles
  - Research Site, Béthune
  - Research Site, Béziers
  - Research Site, Biarritz
  - Research Site, Blaye
  - Research Site, Blois
  - Research Site, Bois-Colombes
  - Research Site, Bois-Guillaume
  - Research Site, Bonneuil-sur-Marne
  - Research Site, Bordeaux
  - Research Site, Boulogne-Billancourt
  - Research Site, Bourges
  - Research Site, Bressuire
  - Research Site, Brest
  - Research Site, Brignoles
  - Research Site, Brive-la-Gaillarde
  - Research Site, Bruay-la-Buissière
  - Research Site, Brunoy
  - Research Site, Cachan
  - Research Site, Caen
  - Research Site, Cagnes-sur-Mer
  - Research Site, Cambrai
  - Research Site, Cannes
  - Research Site, Carcassonne
  - Research Site, Carpentras
  - Research Site, Carquejon
  - Research Site, Castanet-Tolosan
  - Research Site, Castelnau-le-Lez
  - Research Site, Castelnaudary
  - Research Site, Castelsarrasin
  - Research Site, Castres
  - Research Site, Cavaillon
  - Research Site, Cergy
  - Research Site, Chalon-sur-Saône
  - Research Site, Chamalières
  - Research Site, Chambéry
  - Research Site, Champigny-sur-Marne
  - Research Site, Charleville-Mézières
  - Research Site, Chatou
  - Research Site, Château-d'Olonne
  - Research Site, Château-Thierry
  - Research Site, Châteaubernard
  - Research Site, Châteaubriant
  - Research Site, Châtillon-sur-Seine
  - Research Site, Chelles
  - Research Site, Clermont-Ferrand
  - Research Site, Clichy
  - Research Site, Cogolin
  - Research Site, Colmar
  - Research Site, Colombes
  - Research Site, Compiègne
  - Research Site, Condé-sur-l'Escaut
  - Research Site, Conflans STE Honorine
  - Research Site, Coudekerque-Branche
  - Research Site, Courbevoie
  - Research Site, Cournon-d'Auvergne
  - Research Site, Coutances
  - Research Site, Craponne
  - Research Site, Creil
  - Research Site, Crépy-en-Valois
  - Research Site, Créteil
  - Research Site, Croix
  - Research Site, Cusset
  - Research Site, Dax
  - Research Site, Deauville
  - Research Site, Dijon
  - Research Site, Dinan
  - Research Site, Doingt Flamicourt
  - Research Site, Dole
  - Research Site, Douai
  - Research Site, Draguignan
  - Research Site, Drancy
  - Research Site, Dreux
  - Research Site, Dunkirk
  - Research Site, Elbeuf
  - Research Site, Enghien-les-Bains
  - Research Site, Erstein
  - Research Site, Échirolles
  - Research Site, Écully
  - Research Site, Épernay
  - Research Site, Épinal
  - Research Site, Épinay-sur-Seine
  - Research Site, Étampes
  - Research Site, Évecquemont
  - Research Site, Évreux
  - Research Site, Faches-Thumesnil
  - Research Site, Firminy
  - Research Site, Floirac
  - Research Site, Fontainebleau
  - Research Site, Fontenay-sous-Bois
  - Research Site, Forbach
  - Research Site, Fougères
  - Research Site, Fourmies
  - Research Site, Gagny
  - Research Site, Garches
  - Research Site, Gasville-Oisème
  - Research Site, Gennevilliers
  - Research Site, Gentilly
  - Research Site, Givet
  - Research Site, Gleizé
  - Research Site, Gray
  - Research Site, Grenoble
  - Research Site, Grésy-sur-Aix
  - Research Site, Guilherand-Granges
  - Research Site, Guingamp
  - Research Site, Hagondange
  - Research Site, Haguenau
  - Research Site, Hazebrouck
  - Research Site, Hesdin
  - Research Site, Héricourt
  - Research Site, Houilles
  - Research Site, Hyères
  - Research Site, Issoire
  - Research Site, Issy-les-Moulineaux
  - Research Site, Jarville-la-Malgrange
  - Research Site, Juan-les-Pins
  - Research Site, L'Haÿ-les-Roses
  - Research Site, L'Île-Rousse
  - Research Site, La Baule-Escoublac
  - Research Site, La Celle-Saint-Cloud
  - Research Site, La Chaussée-Saint-Victor
  - Research Site, La Ciotat
  - Research Site, La Côte-Saint-André
  - Research Site, La Flèche
  - Research Site, La Garenne-Colombes
  - Research Site, La Madeleine
  - Research Site, La Rochelle
  - Research Site, La Seyne-sur-Mer
  - Research Site, La Varenne-Saint-Hilaire
  - Research Site, La Verpillière
  - Research Site, Lamballe
  - Research Site, Landerneau
  - Research Site, Lanester
  - Research Site, Langon
  - Research Site, Lannemezan
  - Research Site, Lavaur
  - Research Site, Le Blanc-Mesnil
  - Research Site, LE Golfe JUAN
  - Research Site, Le Mans
  - Research Site, Le Pont-de-Beauvoisin
  - Research Site, Le Pontet
  - Research Site, Lens
  - Research Site, Les Sables-d'Olonne
  - Research Site, Les Ulis
  - Research Site, Lesparre-Médoc
  - Research Site, Levallois-Perret
  - Research Site, Liévin
  - Research Site, Lille
  - Research Site, Limoges
  - Research Site, Limoux
  - Research Site, Lisieux
  - Research Site, LIsle-dEspagnac
  - Research Site, Lomme
  - Research Site, Longjumeau
  - Research Site, Loos
  - Research Site, Lorient
  - Research Site, Lunel
  - Research Site, Lyon
  - Research Site, Mainvilliers
  - Research Site, Maisons-Alfort
  - Research Site, Manosque
  - Research Site, Marcq-en-Barœul
  - Research Site, Margency
  - Research Site, Marmande
  - Research Site, Maromme
  - Research Site, Marseille
  - Research Site, Martigues
  - Research Site, Marvejols
  - Research Site, Maubeuge
  - Research Site, Mazamet
  - Research Site, Mende
  - Research Site, Mennecy
  - Research Site, Menton
  - Research Site, Metz
  - Research Site, Millau
  - Research Site, Milly-la-Forêt
  - Research Site, Mons-en-Barœul
  - Research Site, Mont-de-Marsan
  - Research Site, Montargis
  - Research Site, Montauban
  - Research Site, Montbéliard
  - Research Site, Montpellier
  - Research Site, Montreuil
  - Research Site, Montrouge
  - Research Site, Morlaix
  - Research Site, Mouans-Sartoux
  - Research Site, Mulhouse
  - Research Site, Muret
  - Research Site, Nancy
  - Research Site, Nanterre
  - Research Site, Nantes
  - Research Site, Narbonne
  - Research Site, Neufchâteau
  - Research Site, Neuilly-sur-Seine
  - Research Site, Neuves-Maisons
  - Research Site, Nevers
  - Research Site, Nice
  - Research Site, Niort
  - Research Site, Nîmes
  - Research Site, Noisy-le-Grand
  - Research Site, Nœux-les-Mines
  - Research Site, Obernai
  - Research Site, Ollioules
  - Research Site, Orange
  - Research Site, Orléans
  - Research Site, Orly
  - Research Site, Orsay
  - Research Site, Orthez
  - Research Site, Osny
  - Research Site, Oullins
  - Research Site, Ozoir-la-Ferrière
  - Research Site, Pamiers
  - Research Site, Pantin
  - Research Site, Paris
  - Research Site, Pau
  - Research Site, Perpignan
  - Research Site, Pertuis
  - Research Site, Pithiviers
  - Research Site, Plaisance-du-Touch
  - Research Site, Ploemeur
  - Research Site, Ploërmel
  - Research Site, Poissy
  - Research Site, Poitiers
  - Research Site, Pompey
  - Research Site, Pont-à-Mousson
  - Research Site, Pontarlier
  - Research Site, Pontault-Combault
  - Research Site, Pontivy
  - Research Site, Pontoise
  - Research Site, Prades
  - Research Site, Prévessin-Moëns
  - Research Site, Puteaux
  - Research Site, Quimper
  - Research Site, Quincy-sous-Sénart
  - Research Site, Rambouillet
  - Research Site, Reims
  - Research Site, Remiremont
  - Research Site, Rennes
  - Research Site, Revel
  - Research Site, Rezé
  - Research Site, Rillieux-la-Pape
  - Research Site, Roanne
  - Research Site, Rochefort
  - Research Site, Rodez
  - Research Site, Roissy-en-Brie
  - Research Site, Romans-sur-Isère
  - Research Site, Roubaix
  - Research Site, Rouen
  - Research Site, Royan
  - Research Site, Royat
  - Research Site, Rueil-Malmaison
  - Research Site, Saint-Amand-Montrond
  - Research Site, Saint-André-de-Cubzac
  - Research Site, Saint-André-les-Vergers
  - Research Site, Saint-Avold
  - Research Site, Saint-Brieuc
  - Research Site, Saint-Chamond
  - Research Site, Saint-Dié
  - Research Site, Saint-Doulchard
  - Research Site, Saint-Estève
  - Research Site, Saint-Etienne
  - Research Site, Saint-Flour
  - Research Site, Saint-Fons
  - Research Site, Saint-Germain-en-Laye
  - Research Site, Saint-Gély-du-Fesc
  - Research Site, Saint-Herblain
  - Research Site, Saint-Jean-de-Luz
  - Research Site, Saint-Laurent-de-la-Salanque
  - Research Site, Saint-Laurent-du-Var
  - Research Site, Saint-Lô
  - Research Site, Saint-Martin-Boulogne
  - Research Site, Saint-Martin-d'Aubigny
  - Research Site, Saint-Martin-des-Champs
  - Research Site, Saint-Maur-des-Fossés
  - Research Site, Saint-Médard-en-Jalles
  - Research Site, Saint-Michel-sur-Orge
  - Research Site, Saint-Nazaire
  - Research Site, Saint-Orens-de-Gameville
  - Research Site, Saint-Ouen
  - Research Site, Saint-Ouen-l'Aumône
  - Research Site, Saint-Pierre-des-Corps
  - Research Site, Saint-Pol-de-Léon
  - Research Site, Saint-Pol-sur-Ternoise
  - Research Site, Saint-Priest
  - Research Site, Saint-Quentin
  - Research Site, Saint-Raphaël
  - Research Site, Saint-Renan
  - Research Site, Saint-Yrieix-la-Perche
  - Research Site, Salon-de-Provence
  - Research Site, Sarrebourg
  - Research Site, Sarreguemines
  - Research Site, Savigny-sur-Orge
  - Research Site, Sceaux
  - Research Site, Schiltigheim
  - Research Site, Sedan
  - Research Site, Sète
  - Research Site, Sélestat
  - Research Site, Sigean
  - Research Site, Six-Fours-les-Plages
  - Research Site, Somain
  - Research Site, St-Malo
  - Research Site, St.-Jean
  - Research Site, Stains
  - Research Site, Strasbourg
  - Research Site, Sucy-en-Brie
  - Research Site, Suresnes
  - Research Site, Talence
  - Research Site, Tarascon
  - Research Site, Tarbes
  - Research Site, Taverny
  - Research Site, Ternay
  - Research Site, Thann
  - Research Site, Thiais
  - Research Site, Thionville
  - Research Site, Thouars
  - Research Site, Tonnerre
  - Research Site, Toul
  - Research Site, Toulon
  - Research Site, Toulouse
  - Research Site, Tourcoing
  - Research Site, Tournon-sur-Rhône
  - Research Site, Tours
  - Research Site, Trélazé
  - Research Site, Triel-sur-Seine
  - Research Site, Troyes
  - Research Site, Ussel
  - Research Site, Vaison-la-Romaine
  - Research Site, Valenciennes
  - Research Site, Valognes
  - Research Site, Vandœuvre-lès-Nancy
  - Research Site, Vannes
  - Research Site, Vence
  - Research Site, Verrières-le-Buisson
  - Research Site, Versailles
  - Research Site, Vertou
  - Research Site, Vesoul
  - Research Site, Vichy
  - Research Site, Vierzon
  - Research Site, Ville-d'Avray
  - Research Site, Villecresnes
  - Research Site, Villefranche-de-Rouergue
  - Research Site, Villefranche-sur-Mer
  - Research Site, Villemomble
  - Research Site, Villeneuve Saint Georges CEDE
  - Research Site, Villeneuve-la-Garenne
  - Research Site, Villeneuve-Saint-Georges
  - Research Site, Villepreux
  - Research Site, Villers
  - Research Site, Villeurbanne
  - Research Site, Villiers-le-Bel
  - Research Site, Villiers-sur-Orge
  - Research Site, Vincennes
  - Research Site, Vitré
  - Research Site, Vitry-sur-Seine
  - Research Site, Wattignies
  - Research Site, Yvetot